CLINICAL TRIAL: NCT04589286
Title: Phase II Study of Digital Life Coaching in Multiple Myeloma Patients Undergoing Stem Cell Transplantation
Brief Title: Randomized Study of Digital Life Coaching in Myeloma Patients Undergoing Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202511; NCI-2020-08100 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma; Stem Cell Transplant
Keywords: Digital life coaching; Multiple myeloma; Stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pack Health's Digital Life Coaching (DLC) (Experimental): Participants will receive 16 weeks of access to a trained human life coach employed by Pack Health. Coaches will communicate via phone calls, text messages, emails, and links to web-based Pack Health resources plus the addition of generic wellness-related electronic handouts at the time of each email reminder for participant-reported outcome (PRO) assessments
  Interventions: Behavioral: Pack Health's Digital Life Coaching (DLC); Other: Electronic Handouts
- Quasi-usual care control arm (Active Comparator): Participants will receive usual supportive care for stem cell transplantation plus the addition of generic wellness-related electronic handouts at the time of each email reminder for participant-reported outcome (PRO) assessments
  Interventions: Other: Electronic Handouts

INTERVENTIONS:
Behavioral: Pack Health's Digital Life Coaching (DLC) — Pack Health smartphone-based DLC platform
  Other Names: DLC
  Arms: Pack Health's Digital Life Coaching (DLC)
Other: Electronic Handouts — Generic wellness-related electronic handouts

SUMMARY:
Autologous stem cell transplantation (SCT) is the standard of care for fit multiple myeloma (MM) patients; however, the first 100 days after SCT are marked by extensive life disruptions. We have found a 56% relative increase in the use of high-risk benzodiazepine and Z-class (B/Z) drugs for anxiety and insomnia among MM patients during this period. Digital life coaching (DLC), whereby trained coaches work longitudinally with patients through phone calls and text messages to accomplish personal goals, may be able to target anxiety and insomnia in a more integrative manner. This study will investigate whether peri-SCT DLC can lower B/Z usage and improve patient-reported well-being.

DETAILED DESCRIPTION:
This is a single-center, Phase II randomized study of MM patients comparing 16 weeks of DLC access versus quasi-usual care (quasi-usual because both arms will receive generic wellness-related electronic handouts alongside requests for patient-reported outcome (PRO) assessments).

Primary Objective:

To evaluate DLC's impact on B/Z drug usage (excluding lorazepam prescribed for chemotherapy-induced nausea/vomiting, or CINV)

Secondary Objectives:

1. To evaluate DLC's impact on patient-reported general quality of life every 1-2 weeks
2. To evaluate DLC's impact on patient-reported psychosocial distress every 1-2 weeks
3. To evaluate DLC's impact on patient-reported insomnia every 1-2 weeks

Exploratory Objectives:

1. To explore DLC's impact on rates of communications between patients and their treatment teams
2. To explore DLC's impact on clinical outcomes

Participants may continue study treatment (DLC platform access) for 16 weeks from the time of initiating treatment. Participants will not be contacted by the DLC platform vendor after this point. Patients will be followed up at Day +101 after SCT, corresponding to approximately 3 months after SCT.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of one of the following (all referred to as multiple myeloma (MM) for the purposes of this protocol):

  * Multiple myeloma (ICD-10 code: C90.0)
  * Extramedullary plasmacytoma (ICD-10 code: C90.2)
* Planned receipt of autologous stem cell transplantation (SCT) at University of California, San Francisco (UCSF)

  * Patients undergoing outpatient SCT will be eligible
  * Patients who received chemomobilization will be eligible
* Ability to understand a written informed consent form (ICF) document, and the willingness to sign the ICF document

Exclusion Criteria:

* Age < 18 years
* SCT as salvage therapy
* Patient-assessed lack of sufficient English proficiency
* Lack of ownership of a personal smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison of patients with >=1 benzodiazepine and Z-class (B/Z) prescriptions (versus < 1 B/Z prescriptions) | Up to 6 months
  Proportions of patients with >=1 B/Z prescription versus <1 B/Z prescriptions will be compared between arms using chi-square analyses. Participants will be stratified on B/Z usage over time into 3 groups arms based on B/Z-naïve status (i.e., no B/Z usage at time of study enrollment), baseline psychosocial distress, defined as an National Comprehensive Caner Network (NCCN) Distress Thermometer (DT) score of 4 or higher, and baseline insomnia, defined as a Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance short form (SF) 4 item (4a) standardized score of 57 or higher.
Estimate change in B/Z usage | Up to 6 months
  Estimations or differences in changes over time by study group will be performed via a post-estimation test using one-sided t-tests at each assessment. To control the family wise error rate at alpha level of 0.05, the Bonferroni method will be used.
Number of participants with a missing Patient Reported Outcome Measurement Information System (PROMIS) Global Health (GH) assessment | Up to 6 months
  Sensitivity analyses for missing data will be performed on participants with missing PROMIS Global Health assessments
Number of participants with a missing NCCN Distress Thermometer (DT) assessment | Up to 6 months
  Sensitivity analyses for missing data will be performed on participants with missing NCCN DT Assessments
Number of participants with a missing PROMIS Sleep Disturbance SF-4a inventory | Up to 6 months
  Sensitivity analyses for missing data will be performed on participants with missing PROMIS Sleep Disturbance SF-4a inventories.

SECONDARY OUTCOMES:
Change in PROMIS Global Health (GH) Scale Scores | Up to 6 months
  This 10-item inventory is part of the PROMIS series to assess quality of life (QOL) with item scores ranging from 1 to 5. Raw PROMIS scores will be transformed to T-score metrics to reflect a population mean of 50 and a standard deviation of 10. Among cancer patients, a T-score change of 5 points on any PROMIS inventory is generally considered to be clinically meaningful
Change in NCCN Distress Thermometer (DT) Scores | Up to 6 months
  This single-item inventory uses an analog graphic to allow patients to assess their overall distress with a score range of 0 (no distress) to 10 (extreme distress). A score of 4 or higher to differentiate clinically significant distress.
Change in PROMIS 4-item Sleep Disturbance Short Form (SF-4a) Scores | Up to 6 months
  The PROMIS Sleep Disturbance SF-4a inventory will be used to assess quality of sleep, with item scores ranging from 1 to 5. Raw PROMIS scores will subsequently be transformed to T-score metrics to reflect a population mean of 50 and standard deviation of 10. As validated in a previous study of cancer patients, a PROMIS Sleep Disturbance score of 57 or higher will be defined as insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Banerjee, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No